CLINICAL TRIAL: NCT01251575
Title: A Phase II Study to Assess Immunosuppression With Sirolimus Combined With Cyclosporine (CSP) and Mycophenolate Mofetil (MMF) for Prevention of Acute GVHD After Non-Myeloablative HLA Class I or II Mismatched Donor Hematopoietic Cell Transplantation- A Multi-Center Trial
Brief Title: Sirolimus, Cyclosporine, and Mycophenolate Mofetil in Preventing Graft-versus-Host Disease in Treating Patients With Blood Cancer Undergoing Donor Peripheral Blood Stem Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2206.00; NCI-2010-02222 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2206.00 (Other: Fred Hutch/University of Washington Cancer Consortium); P01CA018029 (NIH); P30CA015704 (NIH); RG9213055 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2010-11-29; First posted 2010-12-02 (Estimated); Results first posted 2019-12-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-11

CONDITIONS: Adult Acute Lymphoblastic Leukemia; Adult Acute Myeloid Leukemia; Adult Diffuse Large B-Cell Lymphoma; Adult Myelodysplastic Syndrome; Adult Non-Hodgkin Lymphoma; Aggressive Non-Hodgkin Lymphoma; Childhood Acute Lymphoblastic Leukemia; Childhood Acute Myeloid Leukemia; Childhood Diffuse Large B-Cell Lymphoma; Childhood Myelodysplastic Syndrome; Childhood Non-Hodgkin Lymphoma; Chronic Lymphocytic Leukemia; Chronic Lymphocytic Leukemia in Remission; Chronic Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Hematopoietic and Lymphoid Cell Neoplasm; Mantle Cell Lymphoma; Plasma Cell Myeloma; Prolymphocytic Leukemia; Recurrent Chronic Lymphocytic Leukemia; Refractory Chronic Lymphocytic Leukemia; T-Cell Prolymphocytic Leukemia; Waldenstrom Macroglobulinemia; Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Hodgkin Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Lymphoma, Large B-Cell, Diffuse; Anemia, Refractory, with Excess of Blasts; Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Chronic-Phase; Hematologic Neoplasms; Lymphoma, Mantle-Cell; Multiple Myeloma; Leukemia, Prolymphocytic; Leukemia, Prolymphocytic, T-Cell; Waldenstrom Macroglobulinemia; Hodgkin Disease | interventions — Cyclosporine; Cyclosporins; fludarabine phosphate; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation; Sirolimus; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (fludarabine, transplant, immunosuppression) (Experimental): CONDITIONING: Patients receive fludarabine phosphate IV over 30 minutes on days -4 to -2. Patients also undergo total-body irradiation on day 0.
  TRANSPLANTATION: Patients undergo allogeneic peripheral blood stem cell transplantation.
  IMMUNOSUPPRESSION: Patients receive sirolimus PO QD on days -3 to 180 with taper to day 365; cyclosporine PO BID on days -3 to 150 with taper to day 180; and mycophenolate mofetil PO TID on days 0-30 and then BID to day 100 with taper to day 150.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Cyclosporine; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Mycophenolate Mofetil; Procedure: Peripheral Blood Stem Cell Transplantation; Drug: Sirolimus; Radiation: Total-Body Irradiation

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic peripheral blood stem cell transplant
  Other Names: Allogeneic Hematopoietic Cell Transplantation; allogeneic stem cell transplantation; HSC; HSCT
Drug: Cyclosporine — Given PO or IV
  Other Names: 27-400; Ciclosporin; CsA; Cyclosporin; Cyclosporin A; Gengraf; Neoral; OL 27-400; Sandimmun; Sandimmune; SangCya
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mycophenolate Mofetil — Given PO
  Other Names: Cellcept; MMF
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo allogeneic peripheral blood stem cell transplant
  Other Names: PBPC transplantation; PBSCT; Peripheral Blood Progenitor Cell Transplantation; peripheral stem cell support; Peripheral Stem Cell Transplant; peripheral stem cell transplantation
Drug: Sirolimus — Given PO
  Other Names: AY 22989; RAPA; Rapamune; Rapamycin; SILA 9268A; WY-090217
Radiation: Total-Body Irradiation — Undergo total-body irradiation
  Other Names: TOTAL BODY IRRADIATION; Whole-Body Irradiation

SUMMARY:
This phase II trial studies how well sirolimus, cyclosporine and mycophenolate mofetil works in preventing graft-vs-host disease (GVHD) in patients with blood cancer undergoing donor peripheral blood stem cell (PBSC) transplant. Giving chemotherapy and total-body irradiation before a donor peripheral blood stem cell transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving total-body irradiation together with sirolimus, cyclosporine, and mycophenolate mofetil before and after transplant may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether the incidence of acute GVHD grades II-IV can be reduced to less than the historical rate of 70% with the triple-immunosuppressant combination of cyclosporine (CSP)/mycophenolate mofetil (MMF) with sirolimus in human leukocyte antigens (HLA) class I or class II mismatched related or unrelated donor hematopoietic cell transplantation (HCT) using nonmyeloablative conditioning. The evaluation will be carried out separately among class I and class II mismatched patients.

SECONDARY OBJECTIVES:

I. To evaluate the incidence of non-relapse mortality before day 100.

II. To evaluate the incidences of grades III-IV acute GVHD.

OUTLINE:

CONDITIONING: Patients receive fludarabine phosphate intravenously (IV) over 30 minutes on days -4 to -2. Patients also undergo total-body irradiation on day 0.

TRANSPLANTATION: Patients undergo allogeneic peripheral blood stem cell transplantation.

IMMUNOSUPPRESSION: Patients receive sirolimus orally (PO) once daily (QD) on days -3 to 180 with taper to day 365; cyclosporine PO twice daily (BID) on days -3 to 150 with taper to day 180; and mycophenolate mofetil PO thrice daily (TID) on days 0-30 and then BID to day 100 with taper to day 150.

After completion of study treatment, patients are followed up at 6 months and every year thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Ages > 50 years with hematologic malignancies treatable by related or unrelated HCT
* Ages =< 50 years of age with hematologic diseases treatable by allogeneic HCT who through pre-existing medical conditions or prior therapy are considered to be at high risk for regimen related toxicity associated with a high dose transplant (> 40% risk of transplant-related mortality [TRM]); this criterion can include patients with a HCT-comorbidity index (CI) score of >= 1; transplants should be approved for these inclusion criteria by the principal investigators at the collaborating centers and at Fred Hutchinson Cancer Research Center (FHCRC); all children < 12 years must be discussed with the FHCRC principal investigator (PI) prior to registration
* Ages =< 50 years of age with chronic lymphocytic leukemia (CLL)
* Ages =< 50 years of age with hematologic diseases treatable by allogeneic HCT who refuse a high-dose HCT; transplants must be approved for these inclusion criteria by the principal investigators at the collaborating centers and at FHCRC
* Aggressive non-Hodgkin lymphomas (NHL) and other histologies such as diffuse large B cell NHL: not eligible for autologous HCT, not eligible for high-dose allogeneic HCT, or after failed autologous HCT
* Mantle cell NHL: may be treated in first complete remission (CR); (diagnostic lumbar puncture [LP] required pre-transplant)
* Low grade NHL: with < 6 month duration of CR between courses of conventional therapy
* CLL: must have either 1) failed to meet National Cancer Institute (NCI) Working Group criteria for complete or partial response after therapy with a regimen containing fludarabine (FLU) (or another nucleoside analog, e.g. cladribine [2-CDA], pentostatin) or experience disease relapse within 12 months after completing therapy with a regimen containing FLU (or another nucleoside analog); 2) failed FLU-cyclophosphamide (CY)-Rituximab (FCR) combination chemotherapy at any time point; or 3) have "17p deletion" cytogenetic abnormality; patients should have received induction chemotherapy but could be transplanted in first (1st) CR; 4) patients with a diagnosis of CLL (or small lymphocytic lymphoma) that progresses to prolymphocytic leukemia (PLL); or 5) patients with T-cell CLL or PLL
* Hodgkin lymphoma: must have received and failed frontline therapy
* Multiple myeloma: must have received prior chemotherapy; consolidation of chemotherapy by autografting prior to nonmyeloablative HCT is permitted
* Acute myeloid leukemia (AML): must have < 5% marrow blasts at the time of transplant
* Acute lymphocytic leukemia (ALL): must have < 5% marrow blasts at the time of transplant
* Chronic myeloid leukemia (CML): patients in chronic phase 1 (CP1) must have failed or be intolerant of tyrosine kinase inhibitors (TKIs); patients beyond CP1 will be accepted if they have < 5% marrow blasts at time of transplant
* Myelodysplasia (MDS)/myeloproliferative syndrome (MPS): patients must have < 5% marrow blasts at time of transplant
* Waldenstrom's macroglobulinemia: must have failed 2 courses of therapy
* Patients with related or unrelated donors for whom the best available donor is: a) mismatched at antigen level for any single class I locus (HLA-A, -B, -C) +/- an additional class I mismatch at the allele level OR mismatched at the allele level for any 2 class I loci (if typed at the molecular level) OR mismatched at the antigen or allele level for class II loci HLA-DRB1 and/or - DQB1; must be matched for at least one DRB1 allele and one DQB1 allele; b) there is a likelihood of rapid disease progression while HLA typing and results of a preliminary search and the donor pool suggests that a 10/10 HLA-A, B, C, DRB1 and DQB1 matched donor will not be found; c) there is no HLA-A, -B or -C one locus allelic mismatched donor available
* DONOR: Related or unrelated volunteer donors who are mismatched with the recipient within one of the following limitations:

  * Mismatch for one HLA class I antigen with or without an additional mismatch for one HLA-class I allele, but matched for HLA-DRB1 and HLA-DQ, OR
  * Mismatched for two HLA class I alleles, but matched for HLA-DRB1 and HLA-DQ, OR
  * HLA class I HLA-A, -B, -C allele matched donors allowing for any one or two DRB1 and/or DQB1 antigen allele mismatch
* DONOR: HLA-matching must be based on results of high resolution typing at HLA-A, -B, -C, -DRB1, and -DQB
* DONOR: If the patient is homozygous at the mismatch HLA class I locus or II locus, the donor must be heterozygous at that locus and one allele must match the patient (i.e., patient is homozygous A*01:01 and donor is heterozygous A*01:01, A*02:01); this mismatch will be considered a one-antigen mismatch for rejection only
* DONOR: Donors are excluded when preexisting immunoreactivity is identified that would jeopardize donor hematopoietic cell engraftment; this determination is based on the standard practice of the individual institution; the donor should be excluded if any of the flow cytometric B and T cell cytotoxic cross match assays are positive
* DONOR: Only filgrastim (G-CSF) mobilized PBSC only will be permitted as a hematopoietic stem cell (HSC) source on this protocol

Exclusion Criteria:

* Patients for whom the best available donor is mismatched at both HLA class I and class II
* A positive cross-match exists between the donor and recipient
* Patients with rapidly progressive intermediate or high grade NHL
* Patients with a diagnosis of chronic myelomonocytic leukemia (CMML)
* Patients with refractory anemia with excess blasts (RAEB)-2 who have not received myelosuppressive chemotherapy i.e. induction chemotherapy
* Presence of circulating leukemic blasts (in the peripheral blood) detected by standard pathology for patients with AML, ALL or CML
* Presence of >= 5% circulating leukemic blasts (in the peripheral blood) detected by standard pathology for patients with MDS/MPS
* Central nervous system (CNS) involvement with disease refractory to intrathecal chemotherapy
* Fertile men or women unwilling to use contraceptives during and for up to 12 months following treatment
* Female patients who are pregnant or breast-feeding
* Human immunodeficiency virus (HIV) positive patients
* Patients with active non-hematologic malignancies (except non-melanoma skin cancers) or those with non-hematologic malignancies (except non-melanoma skin cancers) who have been rendered with no evidence of disease, but have a greater than 20% chance of having disease recurrence within 5 years; this exclusion does not apply to patients with non-hematologic malignancies that do not require therapy
* Fungal infections with radiological progression after receipt of amphotericin B or active triazole for greater than 1 month
* Patients with active bacterial or fungal infections unresponsive to medical therapy
* Cardiac ejection fraction < 35% (or, if unable to obtain ejection fraction, shortening fraction of < 26%); ejection fraction is required if the patient is > 50 years of age, or history of cardiac disease or anthracycline exposure; patients with a shortening fraction < 26% may be enrolled if approved by a cardiologist
* Corrected diffusion capacity of carbon monoxide (DLCO) < 40%, total lung capacity (TLC) < 40%, forced expiratory volume in one second (FEV1) < 40% and/or receiving supplementary continuous oxygen; if unable to perform complete pulmonary function tests (PFTs), patients will be excluded if their oxygen saturation is < 95% with a formal six-minute walk test (ambulatory oximetry)
* The FHCRC PI of the study must approve of enrollment of all patients with pulmonary nodules
* Patients with clinical or laboratory evidence of liver disease would be evaluated for the cause of liver disease, its clinical severity in terms of liver function, and the degree of portal hypertension; patients will be excluded if they are found to have fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, alcoholic hepatitis, esophageal varices, a history of bleeding esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction evinced by prolongation of the prothrombin time, ascites related to portal hypertension, bridging fibrosis, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin > 3 mg/dL, or symptomatic biliary disease
* Patients with poorly controlled hypertension on multiple antihypertensives
* Karnofsky scores < 60 or Lansky score < 50
* All patients receiving antifungal therapy voriconazole, posaconazole, or fluconazole must have sirolimus reduced according to the Standard Practice Antifungal Therapy Guidelines
* The addition of cytotoxic agents for "cytoreduction" with the exception of tyrosine kinase inhibitors (such as imatinib), cytokine therapy, hydroxyurea, low dose cytarabine, chlorambucil, or Rituxan will not be allowed within three weeks of the initiation of conditioning
* DONOR: Donor (or centers) who will exclusively donate marrow
* DONOR: Donors who are HIV-positive and/or, medical conditions that would result in increased risk for G-CSF mobilization and harvest of PBSC
* DONOR: Patients who are homozygous at the mismatched HLA class I locus or II locus, the donor is excluded if homozygous at the mismatched locus (i.e., patient is homozygous A*01:01 and donor is homozygous A*02:01); this type of mismatch is considered a two-antigen mismatch and is not allowed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2010-12-01 (Actual); Primary Completion 2018-11-23 (Actual); Study Completion 2019-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Sandmaier, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (5):
- United States (4):
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - VA Puget Sound Health Care System, Seattle, Washington
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington
- Rigshospitalet University Hospital, Copenhagen, Denmark

REFERENCES:
- [Derived] Kornblit B, Storer BE, Andersen NS, Maris MB, Chauncey TR, Petersdorf EW, Woolfrey AE, Flowers MED, Storb R, Maloney DG, Sandmaier BM. Sirolimus with CSP and MMF as GVHD prophylaxis for allogeneic transplantation with HLA antigen-mismatched donors. Blood. 2020 Sep 24;136(13):1499-1506. doi: 10.1182/blood.2020005338. PMID 32603426

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Fludarabine, Transplant, Immunosuppression): CONDITIONING: Patients receive fludarabine phosphate IV over 30 minutes on days -4 to -2. Patients also undergo total-body irradiation on day 0.
  TRANSPLANTATION: Patients undergo allogeneic peripheral blood stem cell transplantation.
  IMMUNOSUPPRESSION: Patients receive sirolimus PO QD on days -3 to 180 with taper to day 365; cyclosporine PO BID on days -3 to 150 with taper to day 180; and mycophenolate mofetil PO TID on days 0-30 and then BID to day 100 with taper to day 150.
  Allogeneic Hematopoietic Stem Cell Transplantation: Undergo allogeneic peripheral blood stem cell transplant
  Cyclosporine: Given PO or IV
  Fludarabine Phosphate: Given IV
  Laboratory Biomarker Analysis: Correlative studies
  Mycophenolate Mofetil: Given PO
  Peripheral Blood Stem Cell Transplantation: Undergo allogeneic peripheral blood stem cell transplant
  Sirolimus: Given PO
  Total-Body Irradiation: Undergo total-body irradiation
Period: Overall Study
Arm/Group | Treatment (Fludarabine, Transplant, Immunosuppression)
Started | 77
Completed | 76
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Fludarabine, Transplant, Immunosuppression)
Number analyzed (Participants) | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 45
  >=65 years | 32
Age, Continuous [Median (Full Range); unit: years] | 63.8 [21.8 to 76.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 67
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 3
  White | 65
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 60
  Denmark | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Grade II-IV Acute Graft Versus Host Disease (GVHD)
Description: Number of patients with grades II-IV acute GVHD
  aGVHD Stages
  Skin:
  1. a maculopapular eruption involving < 25% BSA
  2. a maculopapular eruption involving 25 - 50% BSA
  3. generalized erythroderma
  4. generalized erythroderma w/ bullous formation and often w/ desquamation
  Liver:
  1. bilirubin 2.0 - 3.0 mg/100 mL
  2. bilirubin 3 - 5.9 mg/100 mL
  3. bilirubin 6 - 14.9 mg/100 mL
  4. bilirubin > 15 mg/100 mL
  Gut:
  Diarrhea is graded 1 - 4 in severity. Nausea and vomiting and/or anorexia caused by GVHD is assigned as 1 in severity. The severity of gut involvement is assigned to the most severe involvement noted. Patients w/ visible bloody diarrhea are at least stage 2 gut and grade 3 overall.
  aGVHD Grades Grade II: Stage 1 - 2 skin w/ no gut/liver involvement Grade III: Stage 2 - 4 gut involvement and/or stage 2 - 4 liver involvement Grade IV: Pattern and severity of GVHD similar to grade 3 w/ extreme constitutional symptoms or death
Time Frame: 100 days post-transplant
Measure: Count of Participants; unit: Participants
Groups:
- Class I Mismatch: Patients 1) mismatched at antigen level for any single class I locus (HLA-A, -B, -C) +/- an additional class mismatch at the allele level, or 2) mismatched at the allele level for any 2 class I loci.
- Class II Mismatch: Patients mismatched at the antigen or allele level for class II loci HLA-DRB1 and/or DQB1. Must be matched for at least one DRB1 allele and one DQB1 allele.
Arm/Group | Class I Mismatch | Class II Mismatch
Number analyzed (Participants) | 51 | 25
Participants | 15 | 12

2. Secondary Outcome: Number of Non-Relapse Mortalities
Description: Number of patients expired without disease progression/relapse.
Time Frame: 100 days post-transplant
Population: One subject aborted transplant during conditioning and was counted towards accrual but not evaluated with respect to outcome measures.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Fludarabine, Transplant, Immunosuppression)
Number analyzed (Participants) | 76
Participants | 3

3. Secondary Outcome: Number of Patients With Grade III-IV Acute GVHD
Description: Number of patients with grades III-IV acute GVHD
  aGVHD Stages
  Skin:
  1. a maculopapular eruption involving < 25% BSA
  2. a maculopapular eruption involving 25 - 50% BSA
  3. generalized erythroderma
  4. generalized erythroderma w/ bullous formation and often w/ desquamation
  Liver:
  1. bilirubin 2.0 - 3.0 mg/100 mL
  2. bilirubin 3 - 5.9 mg/100 mL
  3. bilirubin 6 - 14.9 mg/100 mL
  4. bilirubin > 15 mg/100 mL
  Gut:
  Diarrhea is graded 1 - 4 in severity. Nausea and vomiting and/or anorexia caused by GVHD is assigned as 1 in severity. The severity of gut involvement is assigned to the most severe involvement noted. Patients w/ visible bloody diarrhea are at least stage 2 gut and grade 3 overall.
  aGVHD Grades Grade II: Stage 1 - 2 skin w/ no gut/liver involvement Grade III: Stage 2 - 4 gut involvement and/or stage 2 - 4 liver involvement Grade IV: Pattern and severity of GVHD similar to grade 3 w/ extreme constitutional symptoms or death
Time Frame: 100 days post-transplant
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Fludarabine, Transplant, Immunosuppression)
Number analyzed (Participants) | 76
Participants | 2

ADVERSE EVENTS:
Time Frame: AEs: From the start of conditioning to 100 Days post-transplant SAEs: From the start of conditioning to 200 Days post-transplant All-Cause Mortality: Conditioning through 1 Year
Arm/Group | Treatment (Fludarabine, Transplant, Immunosuppression)
All-Cause Mortality (participants affected / at risk) | 21/76
Serious Adverse Events (participants affected / at risk) | 0/76
Other Adverse Events (participants affected / at risk) | 25/76
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Fludarabine, Transplant, Immunosuppression) (N=76)
Acute kidney injury (Renal and urinary disorders) | 4 (4)
Ascites (Gastrointestinal disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 3 (3)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 2 (2)
Creatinine increased (Investigations) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Ejection fraction decreased (Investigations) | 1 (1)
Encephalitis infection (Infections and infestations) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Left ventricular systolic dysfunction (Cardiac disorders) | 2 (2)
Lung infection (Infections and infestations) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Paroxysmal atrial tachycardia (Cardiac disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 3 (4)
Small intestine infection (Infections and infestations) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 2 (3)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Typhlitis (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/75/NCT01251575/Prot_SAP_000.pdf